CLINICAL TRIAL: NCT05888948
Title: Effect of Implementation of a Surgical Emergencies Gradation on Postoperative Outcome in Emergency Operating Theatre Patients of the Amiens-Picardy University Hospital
Brief Title: Surgical Emergencies Gradation and Postoperative Outcome
Acronym: BUGRADA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2022_843_0056
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Emergency Surgery; Mortality
Keywords: emergency surgery; gradation; Complication; mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reducing surgical waiting time has been shown to be associated with a reduction in postoperative morbidity and mortality in this type of surgery. The use of a gradation of surgical emergencies makes it possible to prioritise them in an objective, consensual manner and to carry them out within a theoretical expected waiting time relative to the degree of urgency. The investigators hypothesise that exceeding the theoretical expected waiting time relative to the degree of urgency defined by the gradation of surgical emergencies is associated with an increase in postoperative morbidity and mortality in emergency surgery. The objective is to assess the impact on post-operative morbidity and mortality of waiting times exceeding the theoretical expected time by grading the surgical emergencies of patients undergoing emergency surgery.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old.
* Non-cardiac emergency surgery.

Exclusion Criteria:

* Minor patients
* Emergency cardiac surgery
* Patients under guardianship or curators
* Pregnant women
* Patients who object to their personal data being used in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring non-cardiac emergency surgery at the Amiens-Picardie University Hospital will be included. A posteriori grading will be performed according to an institutionally recognised gradation. Each grade is subject to a theoretical maximum time for surgical management. The surgical waiting time and the waiting time exceeding the theoretical expected time of the gradation will be analysed.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Number Post-operative complications | 1 year
Mortality at 1 year | 1 year
Length of stay in intensive care unit | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No